CLINICAL TRIAL: NCT05285553
Title: MiSight 1 Day Post-Approval Study for Effectiveness and Visual Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAS001/BC
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MiSight 1 day (Experimental): MiSight 1 day
  Interventions: Device: MiSight 1 Day
- Proclear 1 day (Active Comparator): Proclear 1 day
  Interventions: Device: Proclear 1 day

INTERVENTIONS:
Device: MiSight 1 Day — Part 1 of the study - subjects will be randomized to wear MiSight 1 Day for three years.
  Arms: MiSight 1 day
Device: Proclear 1 day — Part 1 of the study - subjects will be randomized to wear Proclear 1 day for three years.
  Part 2 of the study - All the subjects will wear Proclear 1 day lenses for one year.
  Arms: Proclear 1 day

SUMMARY:
The purpose of this post-approval study is to confirm the effectiveness of the MiSight 1 Day lens in clinical practices within the US and to assess the stability of the myopia reduction over one-year post-treatment.

DETAILED DESCRIPTION:
This study is a multicenter, parallel-group, controlled, double-masked (subject and investigator), randomized clinical trial with a total duration of four years.

Part 1 of this study will study the effectiveness of MiSight 1 Day in slowing myopia progression over three years in a US population. Subjects in Part 1 will wear MiSight 1 Day lenses or Proclear 1 day lenses.

Part 2 will study the stability of the effectiveness result over a one-year post-treatment period. All subjects in Part 2 will wear Proclear 1 day lenses. Subjects and investigators will remain masked from Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent and Assent have been completed
2. Be between 8 and 12 years of age inclusive at the time of enrollment.
3. Manifest Refraction - Spherical Equivalent Refractive Error (SERE) at baseline between -0.75 D and -4.00 D inclusive (at the corneal plane) in each eye
4. Best-corrected visual acuity by manifest refraction of +0.10 logMAR (20/25 Snellen equivalent) or better in each eye.
5. Anisometropia: ≤ 1.50D SERE.
6. Astigmatism: ≤ 0.75 D
7. Free of ocular disease or abnormalities (including any corneal scar)
8. Currently have good general health.
9. Agree to accept the lens as assigned by the randomization.
10. Be capable of comprehending the nature of the study and be willing and able to adhere to the instructions set forth in this protocol.
11. Ability to comply with study procedures, including high and low (sub-study only) contrast high and low (sub-study only) lighting visual acuity, axial length, and cycloplegic auto-refraction measurements taken for both eyes.
12. Able to maintain the visit schedule.
13. Willingness to participate in the trial for 4 years.
14. Interested in wearing contact lenses for approximately 10 hours per day and 6 days per week.
15. Possesses, or obtains prior to dispensing, wearable and visually functional (20/40 or better) eyeglasses.

Exclusion Criteria:

1. Current or prior use of any pharmaceuticals or other methods for control of myopia, such as bifocals, progressive addition lenses, orthokeratology, atropine, pirenzepine or any other myopia control treatment.
2. Use of any systemic or topical ocular medications or over-the-counter artificial tears which might interfere with contact lens wear, pupil size, accommodation or refractive state, or require the lenses to be removed during the day.
3. Previously worn or currently wears rigid gas permeable contact lenses, including orthokeratology lenses
4. Has any of the following specific contraindications to MiSight 1 Day lenses at Baseline Visit:

   * Acute and subacute inflammation or infection of the anterior chamber of the eye.
   * Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids.
   * Severe insufficiency of lacrimal secretion (dry eyes).
   * Corneal hypoesthesia (reduced corneal sensitivity), if not aphakic.
   * Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
   * Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
   * Any active corneal infection (bacterial, fungal, or viral).
   * If eyes are red or irritated.
   * The patient is unable to follow lens handling and wear regimen or unable to obtain assistance to do so.
5. Has history of:

   * Corneal ulcer, corneal infiltrates, ocular viral or fungal infections or other recurrent ocular infections.
   * Giant papillary conjunctivitis
   * Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses
   * A known allergy to fluorescein, benoxinate, proparacaine or tropicamide.
   * Corneal hypoesthesia (reduced corneal sensitivity)
6. Keratoconus or an irregular cornea.
7. Strabismus or amblyopia.
8. Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2022-06-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean difference in cycloplegic SERE change from baseline | 3 years
  Mean difference in cycloplegic SERE change from baseline; measured with cycloplegic auto-refraction in Diopters
Mean difference in axial length change from baseline | 3 years
  Mean difference in axial length change from baseline between the MiSight 1 Day group and control lens group, measured in millimeters
Mean difference in rate of cycloplegic SERE change - Part 2 study | 1 year
  Mean difference in rate of cycloplegic SERE change between the Part 1 MiSight 1 Day group and the Part 1 control lens group over one-year post-treatment; measured with cycloplegic auto-refraction in Diopters
Mean difference in rate of axial length - Part 2 study | 1 year
  Mean difference in rate of axial length change between the Part 1 MiSight 1 Day group and Part 1 control lens group over one-year post-treatment.

SECONDARY OUTCOMES:
Percentage of subjects with no appreciable myopic progression | 3 years
  Percentage of subjects with no appreciable myopic progression (-0.25D change or less)
Visual symptoms and the effects on activities of daily living | 3 years
  Visual symptoms and the effects on activities of daily living are measured using a validated PRO Measure

CONTACTS AND LOCATIONS:
Overall Officials: William Gleason, OD, Principal Investigator — Foresight Regulatory Strategies, Inc. (FRS)
Locations (30):
- United States (30):
  - University of Alabama School of Optometry, Birmingham, Alabama
  - Marshall B. Ketchum University Southern California College of Optometry, Fullerton, California
  - Vision Solutions Optometry Inc, La Mesa, California
  - Paje Optometric, Santa Ana, California
  - Coan Eye Care and Optical Boutique, Ocoee, Florida
  - West Broward Eyecare Associates, Tamarac, Florida
  - Bright Eyes Family Vision Care, Tampa, Florida
  - SoLo Eye Care & Eyewear Gallery, Chicago, Illinois
  - Illinois College of Optometry, Chicago, Illinois
  - Chicago College of Optometry, Downers Grove, Illinois
  - Carillon Vision Care, Glenview, Illinois
  - Brain Vision Institute, Schaumburg, Illinois
  - Clinical Optics Research Lab at IU School of Optometry, Bloomington, Indiana
  - Kannarr Eye Care, Pittsburg, Kansas
  - New England College of Optometry, Boston, Massachusetts
  - Cornea and Contact Lens Institute, Edina, Minnesota
  - Vision Source EyeCare, Kansas City, Missouri
  - Athens Eye Care, Athens, Ohio
  - Ohio State University, Columbus, Ohio
  - ProCare Vision Center, Inc., Granville, Ohio
  - Miamisburg Vision Care, Miamisburg, Ohio
  - Eye Care Professionals, Powell, Ohio
  - Southern College of Optometry, Memphis, Tennessee
  - Texas State Optical, Beaumont, Texas
  - University of Houston College of Optometry, Houston, Texas
  - Vision One Eyecare, Katy, Texas
  - Lone Star Vision, Plano, Texas
  - Utah Eye Centers, Ogden, Utah
  - Virginia Pediatric Eye Care, Chesapeake, Virginia
  - Factoria Eye Clinic, Bellevue, Washington